CLINICAL TRIAL: NCT04312074
Title: To Investigate the Effect of Central Arterial Stiffness on the Progression of Male Bladder Dysfunction, Nocturia and Lower Urinary Tract Symptoms
Brief Title: Role of PWV on Male LUTS Progression
Status: Terminated | Type: Observational
Why Stopped: No funding
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Fai NG, Professor, Chinese University of Hong Kong
Other Study IDs: CRE-2019.534
Record Dates: First submitted 2020-03-14; First posted 2020-03-18 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: LUTS
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Male lower urinary tract symptoms (LUTS) is exceedingly common in the general population. Stereotypically, male LUTS have long been attributed to the prostate. However, recent attention has been directed to the bladder dysfunction as a cause of LUTS. LUTS also shares has a close relationship with cardiovascular diseases (CVD), diabetes and metabolic syndrome. These problems could lead to various end-organ damages, via diverse mechanisms, with central arterial stiffness (CAS) is one of them. Amongst the abundant methods for the measurement of CAS, brachial-ankle Pulse Wave Velocity (baPWV) has been shown to be a simple and an accurate approach and is widely used clinically.

From investigators' preliminary work, investigators had shown that baPWV is correlated with the baseline voiding function and voided volume. Investigators postulate that CVD and related diseases would increase CAS, which in turn could cause insult to the urinary bladder. Inevitably, it would lead to bladder dysfunction and LUTS. In the wake of this postulation, a study to investigate the relationship of CAS and the progression of male LUTS is proposed.

DETAILED DESCRIPTION:
Male-LUTS are prevalent, cause bother and impair quality of life (QoL). Not only does it adversely affect the quality of life of men, it is also closely interrelated with many substantial salient medical conditions. LUTS is strongly associated with ageing. The perpetual increase in aging population in Hong Kong and globally, will reflect and amount to the associated costs and relentlessly surmounting burden on the management of the condition in the future. In light of this, better understanding and management of male-LUTS is important for this major health issue.

Stereotypically, male LUTS have long been attributed to be secondary to prostatic enlargement and resulting from its obstruction. However, increasingly conflicting evidences have suggested that LUTS are often unrelated to the prostate. In fact, more attention has been directed to the dysfunction of the bladder, the reservoir and pump of the voiding system, could also contribute a significant component of LUTS, in both male and female. Bladder dysfunction includes detrusor overactivity (overactive bladder), detrusor underactivity (underactive bladder), as well as other structural or functional abnormalities of the urinary tract and its surrounding tissues. Moreover, there are also many other non-urological conditions which can account for urinary symptoms, especially nocturia.As a result, the current concept of managing male LUTS, has expanded from focusing on the prostate to the bladder and even taking into account the perspective of the patient's medical and health condition as a whole.

There are numerous postulated mechanisms to explain the relationship between these medical conditions and LUTS, including sympathetic overtone, release of growth factors / proinflammation markers to stimulate prostate growth, vascular damage to bladder, etc. However, most of them were reported by cross-sectional studies from which the underlying mechanism cannot be proven and the cause and effect relationships cannot be established. Hence, the time / dose relationship between the proposed mechanisms and the development or progression of male LUTS cannot be confirmed. As a result, the exact mechanism leading to development or progression of male LUTS in patients with CVD / DM / MS is still uncertain.

From investigators' preliminary work, investigators had shown that baPWV is correlated with the baseline voiding function and voided volume. Investigators postulate that CVD and related diseases would increase CAS, which in turn could cause insult to the urinary bladder. Inevitably, it would lead to bladder dysfunction and LUTS. In the wake of this postulation, a study to investigate the relationship of CAS and the progression of male LUTS is proposed.

The objectives of the study are: to study the effects of central arterial stiffness on the progression of male bladder dysfunction, nocturia, storage symptoms and voiding symptoms and to explore the effects of central arterial stiffness on the development of complication(s) and the need of surgical intervention in male patients with lower urinary tract symptoms.

400 adult male subjects aged between 40 and 80 years old with non-neurogenic LUTS will be recruited for the study. Having fulfilled all inclusion and exclusion criteria, subjects will then undergo a series of investigation, including bladder diary and baPWV assessment. BaPWV will be measured by an automated machine using the oscillometric cuff technique.

Follow-up assessment will then be arranged at first and second year following the recruitment. During their re-assessment, medical record will be reviewed and the same set of assessment, including bladder diary and baPWV, will be repeated. The changes in voiding function and those of treatment modalities will be correlated with the baseline baPWV and other parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adult male subject aged between 40 and 80 years old.
* Able to consent to the study

Exclusion Criteria:

* Have LUTS secondary to urethral stricture, neurogenic bladder or other structural abnormality
* Have known history of prostate cancer or bladder cancer
* Have been using 5α-reductase inhibitors for the management of male LUTS
* Have history of previous lower urinary tract (bladder, prostate, urethra) surgery or scheduled to have upcoming surgery
* Have history of other pelvic surgery that may affect voiding
* Have bladder stones or an active urinary tract infection within 8 weeks prior to recruitment for the study
* Subject is unable to complete questionnaires adopted in the study

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400 adult male subjects aged between 40 and 80 years old with non-neurogenic LUTS will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in maximal voided volume across the two-year follow-up. | Baseline, Year 1, Year 2
  Maximum voided volume was defined as the highest voided volume recorded in bladder diary.

SECONDARY OUTCOMES:
The number of times an individual passes urine during their main sleep period, from the time they have fallen asleep up to the intention to rise from that period. | Baseline, Year 1, Year 2
  It is assessed by the bladder diary
Incidence of symptom progression | Baseline, Year 1, Year 2
  It is assessed by increase in total International Prostate Symptom Scores IPSS) by 4 points from baseline assessment. For IPSS, the total score ranged from 0 to 35. The higher scores mean the symptom is more severe.
Incidence of adverse events related to voiding, including urinary tract infection, retention of urine, obstructive uropathy, bladder stone formation | Baseline, Year 1, Year 2
  It is assessed by medical record
Incidence of non-medical intervention for voiding symptom, including surgery, other minimally invasive therapy for prostate | Baseline, Year 1, Year 2
  It is assessed by medical record
Incidence of adverse events related to cardiovascular system, such as cerebrovascular accident, myocardial infarction | Baseline, Year 1, Year 2
  It is assessed by medical record
Change in medical therapy for BPH | Baseline, Year 1, Year 2
  It is assessed by medical record
Correlation between the changes in baPWV and changes in voided volume | Baseline, Year 1, Year 2
  Change in baPWV is assessed by Vascular function test, change in voided volume is assessed by bladder diary
Correlation between the changes in baPWV and number of nocturia episode. | Baseline, Year 1, Year 2
  Change in baPWV is assessed by Vascular function test, change in voided volume is assessed by bladder diary

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yee CH, Chan CK, Teoh JYC, Chiu PKF, Wong JHM, Chan ESY, Hou SSM, Ng CF. Survey on prevalence of lower urinary tract symptoms in an Asian population. Hong Kong Med J. 2019 Feb;25(1):13-20. doi: 10.12809/hkmj187502. Epub 2019 Jan 18. PMID 30655460
- [Background] Ng CF, Wong A, Li ML, Chan SY, Mak SK, Wong WS. The prevalence of cardiovascular risk factors in male patients who have lower urinary tract symptoms. Hong Kong Med J. 2007 Dec;13(6):421-6. PMID 18057428
- [Background] Bouwman II, Blanker MH, Schouten BW, Bohnen AM, Nijman RJ, van der Heide WK, Bosch JL. Are lower urinary tract symptoms associated with cardiovascular disease in the Dutch general population? Results from the Krimpen study. World J Urol. 2015 May;33(5):669-76. doi: 10.1007/s00345-014-1398-y. Epub 2014 Sep 25. PMID 25253653
- [Background] Gacci M, Corona G, Sebastianelli A, Serni S, De Nunzio C, Maggi M, Vignozzi L, Novara G, McVary KT, Kaplan SA, Gravas S, Chapple C. Male Lower Urinary Tract Symptoms and Cardiovascular Events: A Systematic Review and Meta-analysis. Eur Urol. 2016 Nov;70(5):788-796. doi: 10.1016/j.eururo.2016.07.007. Epub 2016 Jul 20. PMID 27451136
- [Background] Yee CH, Yip JSY, Cheng NMY, Kwan CH, Li KM, Teoh JYC, Chiu PKF, Wong JH, Chan ESY, Chan CK, Hou SSM, Ng CF. The cardiovascular risk factors in men with lower urinary tract symptoms. World J Urol. 2019 Apr;37(4):727-733. doi: 10.1007/s00345-018-2432-2. Epub 2018 Aug 6. PMID 30083830
- [Background] Victor RG, Li N, Blyler CA, Mason OR, Chang LC, Moy NPB, Rashid MA, Weiss JP, Handler J, Brettler JW, Sagisi MB, Rader F, Elashoff RM. Nocturia as an Unrecognized Symptom of Uncontrolled Hypertension in Black Men Aged 35 to 49 Years. J Am Heart Assoc. 2019 Mar 5;8(5):e010794. doi: 10.1161/JAHA.118.010794. PMID 30827133
- [Background] Tsuchikura S, Shoji T, Kimoto E, Shinohara K, Hatsuda S, Koyama H, Emoto M, Nishizawa Y. Brachial-ankle pulse wave velocity as an index of central arterial stiffness. J Atheroscler Thromb. 2010 Jun 30;17(6):658-65. doi: 10.5551/jat.3616. Epub 2010 May 13. PMID 20467192
- [Background] Uzun H, Cicek Y, Kocaman SA, Durakoglugil ME, Zorba OU. Increased pulse-wave velocity and carotid intima-media thickness in patients with lower urinary tract symptoms. Scand J Urol. 2013 Oct;47(5):393-8. doi: 10.3109/21681805.2013.780185. Epub 2013 Mar 26. PMID 23528066
- [Background] Yamaguchi O. Latest treatment for lower urinary tract dysfunction: therapeutic agents and mechanism of action. Int J Urol. 2013 Jan;20(1):28-39. doi: 10.1111/iju.12008. Epub 2012 Nov 28. PMID 23190275
- [Background] Lombardo R, Tubaro A, Burkhard F. Nocturia: The Complex Role of the Heart, Kidneys, and Bladder. Eur Urol Focus. 2020 May 15;6(3):534-536. doi: 10.1016/j.euf.2019.07.007. Epub 2019 Aug 5. PMID 31395515